CLINICAL TRIAL: NCT04389996
Title: COVID-19 Pandemic Impact on Patients With Cancer - a Danish Survey
Acronym: COPICADS
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Stefan Starup Jeppesen, Head of Department of Oncology, Associate professor, PhD, Odense University Hospital
Other Study IDs: OP_1132
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Cancer
Keywords: Cancer; Quality of Life; COVID-19
MeSH Terms: conditions — Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cancer: Survey
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Patients will be sent a survey incl. EORTC QLQ-C30

SUMMARY:
The outbreak of coronavirus was categorized as a global pandemic in March 2020. The Danish government recommends social distancing during the COVID-19 pandemic. Long-term social distancing and fear of disease can lead to anxiety, depression and the feeling of loneliness. All these factors might affect the quality of life (QoL).

The aim of this study is to investigate the overall QoL for patients with cancer during the COVID-19 pandemic with special focus on emotional functioning.

DETAILED DESCRIPTION:
Since the detection of the novel coronavirus also called COVID-19 in December 2019 it has affected many people worldwide. The outbreak of coronavirus was categorized as a global pandemic in March 2020.

The focus of the Danish health care system is on patients infected with COVID-19. In order to limit the spread of this disease, the Danish government recommends social distancing during the COVID-19 pandemic. Unfortunately, long-term social distancing and fear of disease can lead to anxiety, depression and the feeling of loneliness. All these factors might affect the quality of life (QoL). The fear of the COVID-19 among the Danish population is thought to be high since cancer referrals to the departments have decreased markedly during the pandemic - probably because people avoid appointments at the hospital or general practitioner.

A population that may be seriously impacted by the COVID-19 disease is the group of patients with cancer. Patients with cancer are in a high risk of serious illness of infections because the cancer and antineoplastic treatment often weaken the immune system. However, no reports are available regarding higher incidence of COVID-19 in patients with cancer. The patients with cancer might be practicing social distancing even more than the general population and the well-being for this group of patients may be even more affected by the COVID-19 disease.

In Denmark, during the coronavirus outbreak different treatment guidelines have been conducted to minimize the risk of infection with the COVID-19 virus, but also the impact of pandemic on the cancer treatment and follow-up program. Also European recommendations have been conducted to help clinicians deal with various aspects of cancer care. Immunotherapy for patients with cancer can be changed from a 3 week schedule to 6 week schedule and many palliative radiation treatments can be changed from a schedule of 10 fractions to 5 fractions. Furthermore it is recommended by the European societies of medical oncology and radiation oncology to avoid hospital appointments for patients with cancer. In follow-up programmes outpatient clinic visits can be done over the phone or may even be postponed.

Avoiding exposure to the COVID-19 virus can be essential for patients with cancer. The new pandemic situation can cause serious concerns for this group of patients. Many visits at the oncological outpatient clinics are being cancelled or appointments are done by phone to avoid as many contacts to the health system as possible. The lack of face-to-face contact to the staff at the Departments of Oncology might cause worries and anxiety for the patients and their relatives, because of the risk of less detailed information regarding side effects of treatment as well as cancer related symptoms. Patients may also worry that their antineoplastic treatment will be discontinued or changed due to reduction of visits at the outpatient clinics. Overall the QoL can be affected for patients with cancer. A structured and unified approach to COVID-19 prevention and care specific to cancer patients and cancer centers is highly needed. Many of the initiatives to avoid face-to-face contact during the COVID-19 pandemic e.g. telephonic or web-technology contacts for consultation may continue in the time after the COVID-19 pandemic. It is therefore of interest to explore the patients' QoL and to investigate their satisfaction with cancer treatment and follow-up during the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer
* Patients who are receiving cancer treatment or patients in follow-up for a cancer diagnosis
* Age 18+

Exclusion Criteria:

* Patients without "eBoks" - a secure electronic mailbox used to receive digital mail from the private sector

Ages: 18 Years to 125 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited at the Department of Oncology and the Department of Haemotology, Odense University Hospital, Denmark.
  Patients are either receiving cancer treatment or in follow-up for a cancer diagnosis
Sampling Method: Probability Sample
Enrollment: 6810 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Overall Quality of Life | One measurement of EORTC QLQ-C30 and a survey created for the purpose will be performed through study completion, an average of 1 months
  EORTC (European Organisation for Research and Treatment of Cancer) QLQ-C30 (Quality of Life Questionnaire core 30) - The QLQ-C30 is a standardized cancer-specific 30-itemed instrument. Scores are transformed linearly to a zero to 100 scale. A higher score on the functional scale and the global Health related Quality of Life indicates better functioning.
  In the current study, the items addressing global quality of life and health: "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" will be used to get a pure expression of QoL.
  The EORTC QLQ-C30 scores in this study will be compared with QoL for Danish Cancer patients in the period before COVID-19 (https://www.cancer.dk/dyn/resources/File/file/3/8373/1574778638/kraeftens-bekaempelses-barometerundersoegelse-2019.pdf). Results on overall QoL is listed on page 36.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan S Jeppesen, MD, PhD, Principal Investigator — Odense University Hospital
Locations (2):
- Denmark (2):
  - Department of Haemotology, Odense University Hospital, Odense, Region Syddanmark
  - Department of Oncology, Odense University Hospital, Odense C

IPD SHARING:
Plan to Share IPD: Undecided